CLINICAL TRIAL: NCT06548711
Title: Director of Oncology Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Brief Title: Effect of Transcutaneous Acupoint Electrical Stimulation (TAES) on Postoperative Cough in Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kong Fanming (Other)
Responsible Party: Sponsor-Investigator, Kong Fanming, Director of Oncology Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYLL2024[Z]026
Record Dates: First submitted 2024-07-29; First posted 2024-08-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Cough; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Due to the specific nature of acupuncture clinical research, it is difficult to accomplish double blinding of subjects and operators, so this trial was blinded to subjects and statisticians only. The statistical analyst was a non-subject and was not aware of the patient treatment or the trial protocol. For all patients who participated in acupuncture, blinded evaluation questions were asked at the 1 week after acupuncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAS group (Experimental): The patient takes a sitting position, uses alcohol to wipe the skin at the selected acupoint, waits for it to dry, and then applies the electrode patch. Connect the percutaneous acupoint electric stimulator and provide transcutaneous acupoint electric stimulation, selecting a continuous wave at 2 Hz.
  Interventions: Other: Transcutaneous Acupoint Electrical Stimulation (TAES)
- Sham TEAS group (Sham Comparator): The electrode patch is placed on the acupoint, similar to the TEAS group patients, but without starting the electric stimulation, and indicates to the patient that there will be no special sensation during the treatment process. The electrode is well protected during the operation and will not come off.
  Interventions: Other: Transcutaneous Acupoint Electrical Stimulation (TAES)

INTERVENTIONS:
Other: Transcutaneous Acupoint Electrical Stimulation (TAES) — Transcutaneous acupoint electrical stimulation (TAES) is a non-invasive treatment method that delivers gentle electrical pulses through the skin to specific acupuncture points on the body. This technique aims to mimic the effects of traditional acupuncture, providing a convenient and painless method of treatment.

SUMMARY:
Observation and exploration of the improvement in cough symptoms in postoperative lung cancer patients with Transcutaneous Acupoint Electrical Stimulation (TAES), the change in Cough Symptom Score (CSS) compared to baseline, the change in Visual Analog Scale (VAS) score for cough symptoms compared to baseline, the change in total score of Leicester Cough Questionnaire-Mandarin Chinese version (LCQ-MC) compared to baseline, and overall evaluation of treatment effectiveness by patients. A total of 84 postoperative lung cancer patients with cough were strictly selected according to the inclusion/exclusion criteria and treated and followed up according to the research plan requirements. Clinical observation forms were completed and clinical data were recorded in the database. Statistical analysis was performed on relevant clinical observation indicators to report research results and write related papers.

DETAILED DESCRIPTION:
To obtain sufficient evidence from evidence-based medicine, prospective, random, blind, and controlled clinical trials are adopted to evaluate the effectiveness and safety of TEAS in treating postoperative cough in lung cancer patients. This study aims to provide a potential non-pharmacological treatment option for postoperative cough patients with lung cancer, improve the quality of life of postoperative lung cancer patients, identify the population that is more likely to benefit from TEAS treatment and provide a solid scientific basis and guidance for personalized acupuncture treatment for postoperative cough in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old - Surgery performed under general anesthesia for radical resection of lung cancer or lung cancer resection combined with lymph node dissection.
* Pathological confirmation of primary lung cancer after surgery.
* Duration of persistent dry cough after lung surgery ≥2 weeks.
* Consciousness, ability to express opinions clearly, and voluntary signing of informed consent.

Exclusion Criteria:

* Patients diagnosed with acute respiratory system diseases within 1 month.
* Patients diagnosed with pneumonia based on chest X-ray.
* Patients with a history of asthma or tuberculosis.
* Patients with uncontrolled hyperthyroidism, severe hypertension, heart disease, systemic infection, coagulation disorders (hypercoagulable state or bleeding tendency), or other severe systemic diseases.
* Patients who have used steroid drugs within the past 3 months.
* Patients who have taken angiotensin-converting enzyme inhibitors (ACEIs) within the past 6 months.
* Patients with surgical incisions, skin allergies, wounds, or infections in the treatment area.
* Patients who cannot tolerate transcutaneous acupoint electrical stimulation or withdraw during the procedure.
* Patients with contraindications to transcutaneous electrical stimulation or implanted electrophysiological devices.
* Patients who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
LCQ-MC | Prior to treatment (baseline), at the end of treatment (week 2), and 2 weeks after the end of treatment (week 4)
  The questionnaire consists of 19 items, each of which is divided into 7 levels according to the severity, including the impact of chronic cough on the physiological domain (chest pain, cough, sputum, fatigue, sleep, hoarseness, etc.), psychological domain (feeling embarrassed, anxious, depressed, annoyed, etc.), and social domain (work, daily life, leisure activities, conversation, phone calls, interference with friends or family members). The score for each domain is the total score of each item in that domain divided by the number of questions (scored from 1 to 7), and the total score is the sum of the scores for the three domains (scored from 3 to 21). A higher score represents a better patient's health condition.

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No